CLINICAL TRIAL: NCT07036328
Title: Transcranial Magnetic Stimulation (TMS) to Slow Down Cognitive Decline in Alzheimer's Disease (AD): TMSLA - a Monocentric Randomized Controlled Trial.
Brief Title: Transcranial Magnetic Stimulation to Slow Down Cognitive Decline in Alzheimer's Disease
Acronym: TMSLA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Willem de Haan (Other)
Responsible Party: Sponsor-Investigator, Willem de Haan, Principal Investigator, Amsterdam UMC, location VUmc
Organization: Amsterdam UMC, location VUmc (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2024.0870
Record Dates: First submitted 2025-04-24; First posted 2025-06-25 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-05

CONDITIONS: Alzheimer Disease; Alzheimer Disease, Early Onset
MeSH Terms: conditions — Alzheimer Disease | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Verum (Experimental): Verum rTMS
  Interventions: Device: repetitive transcranial magnetic stimulation
- Sham (Sham Comparator): sham rTMS
  Interventions: Device: sham repetitive transcranial magnetic stimulation

INTERVENTIONS:
Device: repetitive transcranial magnetic stimulation — 20 Hz repetitive transcranial magnetic stimulation targeted at the precuneus
  Arms: Verum
Device: sham repetitive transcranial magnetic stimulation — 20 Hz sham repetitive transcranial magnetic stimulation targeted at the precuneus
  Arms: Sham

SUMMARY:
New amyloid-targeting drugs for Alzheimer's disease (AD) offer minimal or unclear efficacy and often cause adverse events, highlighting the need for new therapies. In recent years, repetitive transcranial magnetic stimulation (rTMS) has shown increasing success. A recent randomized, double-blind, sham-controlled, phase 2 demonstrated promising results from a 24-week rTMS treatment protocol targeting the precuneus. This brain region is considered a main hub of the human brain connectome and a prominent area of AD pathology. The results showed stable cognitive performance and increased brain activity in the treatment group, whereas the sham group worsened. A replication study is planned to further investigate the working mechanism of precuneus-rTMS in AD and to improve understanding of its therapeutic potential.

ELIGIBILITY:
Inclusion Criteria:

* Biomarker-supported Alzheimer's disease (abnormal CSF p-tau/Aβ42 ratio of > 0.023 or amyloid PET positive).
* Between 50 and 85 years old.
* Clinical Dementia Rating (CDR) score of 0.5 or 1.
* Mini-Mental State Examination (MMSE) score between 18 and 26.
* Presence of a caregiver.

Exclusion Criteria:

* Medical history of neurodegenerative diseases other than AD, stroke, or epilepsy.
* Severe psychiatric dysregulation, hampering successful study participation and leading to possible cognitive impairment. Eligibility for participation will be based on clinical evaluation by an expert neurologist and/or psychiatrist.
* Extensive cerebrovascular damage on MRI classified as Fazekas level 2 or 3. Patients with abnormalities classified as Fazekas level 3 are excluded. For Fazekas level 2, patient's eligibility for participation will be evaluated by an expert neurologist.
* Presence of metal in the head or cranial/thoracic implants, including cochlear implants.
* Cholinesterase inhibitors with unstable dosage in the last 2 months.
* Extreme claustrophobia or metallic objects in or on the body, preventing MRI and MEG examination.
* Previous rTMS treatment (for blinding reasons).

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2025-04-07 (Actual); Primary Completion 2028-01 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
CDR - Sum of Boxes | from enrollment to 3 month follow-up
  Clinical dementia rating - sum of boxes

SECONDARY OUTCOMES:
Magnetoencephalography (MEG): Spectral analysis | from baseline to week 24 (post-treatment)
  Power spectral density (µV²/Hz) computed for different frequency bands .
Cerebrospinal fluid (CSF) biomarkers | from baseline to week 24 (post-treatment)
  Cerebrospinal fluid (CSF) biomarkers are typically reported in picograms per milliliter (pg/mL). This applies to:
  Amyloid-beta (Aβ₁-₄₂): pg/mL Total tau (t-tau): pg/mL Phosphorylated tau (p-tau, e.g., p-tau181): pg/mL
Neuropsychological evaluation: Trail Making Test | from baseline to week 24 (post-treatment)
  Assesses visual attention, processing speed, and task switching. Unit: Seconds (completion time)
Amsterdam instrumental activities of daily living questionnaire (AmsterdamiADL); | baseline to 3 month follow-up
  The Amsterdam Instrumental Activities of Daily Living (A-IADL) Questionnaire is a validated tool that assesses cognitive functioning through everyday tasks, with scores ranging from approximately 20 (severe impairment) to 70 (no impairment).
Mini mental state examination (MMSE) | baseline to 3-month follow up.
  The mini-mental state examination (MMSE) test is a 30-point questionnaire that is used extensively in clinical and research settings to measure cognitive impairment. Higher is better.
Neuropsychiatric Inventory Questionnaire (NPI-Q) | baseline to 3 month follow up
  The Neuropsychiatric Inventory Questionnaire (NPI-Q) is a brief, informant-based tool that assesses 12 neuropsychiatric symptoms in dementia, with total severity scores ranging from 0 to 36 and distress scores from 0 to 60.
Quick Inventory of Depressive Symptomatology (QIDS) | baseline to 3-month follow up
  The Quick Inventory of Depressive Symptomatology (QIDS) is a clinician-rated tool that measures the severity of depressive symptoms, with total scores ranging from 0 (no depression) to 27 (severe depression).
Magnetoencephalography (MEG): Corrected Amplitude Envelope Correlation (AEC-c) | From baseline to week 24 (post-treatment)
  Correlation of the amplitude envelopes of band-pass filtered signals, corrected for signal leakage.
Magnetoencephalography (MEG): Phase Lag Index (PLI) | baseline to week 24 (post-treatment)
  A measure of phase synchronization that is robust to volume conduction.
Magnetoencephalography (MEG): Joint Permutation Entropy (JPE) | baseline to week 24 (post-treatment)
  A nonlinear measure of signal complexity and diversity in joint time series.
Neuropsychological evaluation: Verbal Fluency Test | baseline to week 24 (post-treatment)
  Measures verbal production and executive functioning.
  Phonemic fluency (letters D, A, T) Unit: Number of words per 1 minute
  Semantic fluency (animals) Unit: Number of words per 1 minute
Neuropsychological evaluation: Visual Association Test (VAT) | baseline to week 24 (post-treatment)
  Detects signs of anterograde amnesia through object-pair associations. Unit: Number of correct associations (maximum score: 12)
Neuropsychological evaluation: Stroop Color and Word Test | baseline to week 24 (post-treament)
  Evaluates cognitive flexibility, inhibition, and processing speed. Unit: Seconds (per condition), Errors (count)
Neuropsychological evaluation: WAIS-III Digit Span (Forward and Backward) | baseline to week 24 (post-treatment)
  Assesses attention and verbal working memory. Unit: Span length (maximum correctly repeated digit sequences)
Neuropsychological evaluation: Rey Auditory Verbal Learning Test (RAVLT) | baseling to week 24 (post-treatment)
  Evaluates verbal learning and declarative memory.
  Immediate recall (Trials I-V) Unit: Total number of words recalled
  Delayed recall Unit: Number of words recalled
  Recognition Unit: Number of correct recognitions

CONTACTS AND LOCATIONS:
Locations (1):
- Amsterdam UMC, Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
The individual participant data will be made available upon reasonable request to the corresponding author in consultation with the data protection officer
Time Frame: Data will be shared after the study completion indefinitely
Access Criteria: Upon reasonable request

REFERENCES:
- [Background] Koch G, Casula EP, Bonni S, Borghi I, Assogna M, Minei M, Pellicciari MC, Motta C, D'Acunto A, Porrazzini F, Maiella M, Ferrari C, Caltagirone C, Santarnecchi E, Bozzali M, Martorana A. Precuneus magnetic stimulation for Alzheimer's disease: a randomized, sham-controlled trial. Brain. 2022 Nov 21;145(11):3776-3786. doi: 10.1093/brain/awac285. PMID 36281767